CLINICAL TRIAL: NCT05062759
Title: A Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled, Phase 3b Study to Evaluate the Potential Effect of Tezepelumab on the Humoral Immune Response to Seasonal Quadrivalent Influenza Vaccination in Adolescent and Young Adult Participants With Moderate to Severe Asthma (VECTOR)
Brief Title: Study to Assess the Effect of Tezepelumab on the Immune Response to Influenza Vaccination in Participants With Asthma
Acronym: VECTOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5180C00031
Record Dates: First submitted 2021-08-23; First posted 2021-09-30 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Moderate to Severe Asthma
Keywords: Tezepelumab; Humoral Immune Response; Quadrivalent Influenza Vaccination; Antibody response; Subcutaneous
MeSH Terms: interventions — tezepelumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Neither the participant nor any of the investigators or sponsor staff who are involved in the treatment or clinical evaluation and monitoring of the participants will be aware of the treatment received. Since tezepelumab and placebo are not visually distinct, study intervention will be handled by a qualified person (eg, pharmacist or study nurse) at the site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tezepelumab (Experimental): Participants will be randomized to receive tezepelumab 210 mg administered at Weeks 0, 4, 8 and 12. Participants will also receive a single dose of inactivated quadrivalent seasonal influenza vaccine intramuscularly at Week 12, prior to the fourth dose of study intervention.
  Interventions: Drug: Tezepelumab
- Placebo to Tezepelumab (Placebo Comparator): Participants will be randomized to receive placebo SC Q4W, administered at Weeks 0, 4, 8 and 12. Participants will also receive a single dose of inactivated quadrivalent seasonal influenza vaccine intramuscularly at Week 12, prior to the fourth dose of study intervention.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tezepelumab — 210 mg SC injection Q4W.
  Arms: Tezepelumab
Drug: Placebo — SC injection Q4W.
  Arms: Placebo to Tezepelumab

SUMMARY:
This is a Phase 3b, multicenter, randomized, double-blind, parallel group, placebo-controlled study designed to investigate the potential effect of tezepelumab (210 mg subcutaneous [SC] every 4 weeks [Q4W]) on antibody responses following seasonal quadrivalent influenza virus vaccination in the fall/winter 2021-2022 in the USA.

DETAILED DESCRIPTION:
Participants with moderate to severe asthma will enter the screening period of a minimum of 2 weeks to allow adequate time for all of the eligibility criteria to be evaluated. They will be randomized 1:1 to receive tezepelumab 210 mg or placebo SC Q4W, administered at Weeks 0, 4, 8 and 12. Randomization will be monitored to ensure at least 50% of the randomized participants are between the ages of 12 to 17 years.

Participants will receive a single dose of inactivated quadrivalent seasonal influenza vaccine intramuscularly at Week 12, prior to the fourth dose of study intervention.

Serum samples for evaluation of antibody response will be drawn at Week 12 (pre-vaccination) and at Week 16 (4 weeks post-vaccination) when humoral response to the vaccination is expected to be fully developed.

The End of Treatment (EOT) Visit will be conducted at Week 16 and a final Follow-up Visit and the End of Study Visit will be conducted at Week 28.

ELIGIBILITY:
Inclusion Criteria:

* Documented physician-diagnosed asthma for at least 12 months prior to Visit 1.
* Morning pre-bronchodilator FEV1 (Forced expiratory volume) of > 50% predicted normal value at Visit 1 or Visit 2.
* Body weight ≥ 40 kg.
* For women of childbearing potential, a negative urine pregnancy test is required prior to administration of study intervention at Visit 3.
* Must have 'not well-controlled' asthma.

Exclusion Criteria:

* Clinically important pulmonary disease other than asthma.
* Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physical impairment.
* Life-threatening asthma
* History of cancer.
* Allergy to eggs, if egg based influenza vaccine will be administered.
* History of anaphylaxis to any biologic therapy.
* Current smokers or participants with smoking history ≥ 10 pack-years and participants using vaping products, including electronic cigarettes. Former smokers with a smoking history of < 10 pack-years and users of vaping or e-cigarette products must have stopped for at least 6 months prior to Visit 1 to be eligible.
* History of alcohol or drug abuse within 12 months prior to the date of informed consent.
* Major surgery within 8 weeks prior to Visit 1 or planned surgical procedures during the conduct of the study.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-07-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Research Site, Bakersfield, California
  - Research Site, Huntington Beach, California
  - Research Site, Miami, Florida
  - Research Site, Columbia, Missouri
  - Research Site, Northfield, New Jersey
  - Research Site, Dayton, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tyler, Texas
  - Research Site, Waco, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at:
  https://astrazenecagrouptrials.pharmacm.com /ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Cole J, Capala-Szczurko I, Roseti S, Chen C, Caveney S, Aksyuk AA, Streicher K, Ponnarambil S, Colice G. Effect of Tezepelumab on the Humoral Immune Response to Seasonal Quadrivalent Influenza Vaccination in Patients with Moderate to Severe Asthma: The Phase 3b VECTOR Study. Pulm Ther. 2024 Mar;10(1):53-67. doi: 10.1007/s41030-023-00245-9. Epub 2023 Dec 8. PMID 38064153
- See also: CSR Synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5180C00031&attachmentIdentifier=30f0d69f-126e-4f79-8bc8-0542f713c2b0&fileName=D5180C00031_CSR_Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 15 study centres in the United States between 23 August 2021 and 18 July 2022.
Pre-assignment Details: The Screening period was 2 to 3 weeks before randomisation. Patients were randomised in a 1:1 ratio to receive tezepelumab or placebo. All the study assessments were performed as per the Schedule of Activities.
Groups:
- Tezepelumab: Patients received at least 1 injection of tezepelumab 210 mg administered subcutaneously every 4 weeks by APFS
- Placebo: Patients received at least 1 injection of placebo administered subcutaneously every 4 weeks by APFS
Period: Overall Study
Arm/Group | Tezepelumab | Placebo
Started | 35 | 35
Completed | 34 | 34
Not Completed | 1 | 1
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: All patients randomised and receiving any study intervention were included in the Full analysis set, irrespective of their CSP adherence and continued participation in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tezepelumab | Placebo | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.3 (2.3) | 16.6 (3.1) | 16.5 (3.0)
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0
  Children (2-11 years) | 0 | 0 | 0
  Adolescents (12-17 years) | 22 | 21 | 43
  Adults (18-64 years) | 13 | 14 | 27
  From 65-84 years | 0 | 0 | 0
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 21 | 24 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 18
  Not Hispanic or Latino | 27 | 25 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 24 | 23 | 47
  Black or African American | 8 | 12 | 20
  Asian | 1 | 0 | 1
  American Indian or Alaska Native | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Post-vaccination Strain-specific Hemagglutination Inhibition (HAI) Antibody Geometric Mean Fold Rises (GMFRs)
Description: Effect of tezepelumab on the humoral immune response following seasonal influenza virus vaccination in adolescent and young adult participants with moderate to severe asthma was assessed.
  HAI assay was not performed for H3N2 strain due to the known low haemagglutination effect.
Time Frame: From Week 12 to Week 16
Population: Vaccine immunogenicity analysis set consisted of all randomised patients who received the influenza vaccine plus at least 1 dose of tezepelumab or placebo, had pre and post vaccination HAI or Microneutralization antibody measurements, had no influenza infection prior to Visit 7 (Week 16), and had no protocol deviation, judged to have the potential to interfere with the generation or interpretation of an antibody response.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fold change
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 33 | 33
Fold change
  Influenza A H1N1 | 7.34 (1.361) [lower limit 1.361] | 4.75 (1.455) [lower limit 1.455]
  Influenza B Yamagata Lineage | 1.76 (0.955) [lower limit 0.955] | 1.46 (0.937) [lower limit 0.937]
  Influenza B Victoria Lineage | 2.94 (1.054) [lower limit 1.054] | 2.90 (0.841) [lower limit 0.841]
Statistical Analysis 1: Comparison: Tezepelumab vs Placebo; Influenza A H1N1 Ratio of placebo over tezepelumab. Results based on ANCOVA model; Test type: Other; Geometric Least square (LS) mean ratio = 0.65, 90% CI 2-sided [0.43 to 0.98]
Statistical Analysis 2: Comparison: Tezepelumab vs Placebo; Influenza B Yamagata Lineage Ratio of placebo over tezepelumab. Results based on ANCOVA model; Test type: Other; Geometeric LS mean ratio = 0.83, 90% CI 2-sided [0.60 to 1.15]
Statistical Analysis 3: Comparison: Tezepelumab vs Placebo; Influenza B Victoria Lineage Ratio of placebo over tezepelumab. Results based on ANCOVA model; Test type: Other; Geometric LS mean ratio = 0.99, 90% CI 2-sided [0.71 to 1.37]

2. Primary Outcome: Post-vaccination Strain-specific Microneutralization (MN) Antibody GMFRs
Description: Effect of tezepelumab on the humoral immune response following seasonal influenza virus vaccination in adolescent and young adult participants with moderate to severe asthma was assessed.
Time Frame: From Week 12 to Week 16
Population: Vaccine immunogenicity analysis set consisted of all randomised patients who received the influenza vaccine plus at least 1 dose of tezepelumab or placebo, had pre and post vaccination HAI or MN antibody measurements, had no influenza infection prior to Visit 7 (Week 16), and had no protocol deviation, judged to have the potential to interfere with the generation or interpretation of an antibody response.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fold change
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 33 | 33
Fold change
  Influenza A H1N1 | 14.56 (2.581) [lower limit 2.581] | 10.62 (2.409) [lower limit 2.409]
  Influenza A H3N2 | 4.73 (1.509) [lower limit 1.509] | 5.90 (3.180) [lower limit 3.180]
  Influenza B Yamagata Lineage | 4.00 (1.541) [lower limit 1.541] | 3.56 (2.206) [lower limit 2.206]
  Influenza B Victoria Lineage | 4.08 (2.279) [lower limit 2.279] | 5.04 (1.723) [lower limit 1.723]
Statistical Analysis 1: Comparison: Tezepelumab vs Placebo; Influenza A H1N1 Ratio of placebo over tezepelumab. Results based on ANCOVA model; Test type: Other; Geometeric LS mean ratio = 0.73, 90% CI 2-sided [0.42 to 1.28]
Statistical Analysis 2: Comparison: Tezepelumab vs Placebo; Influenza A H3N2 Ratio of placebo over tezepelumab. Results based on ANCOVA model; Test type: Other; Geometeric LS mean ratio = 1.25, 90% CI 2-sided [0.72 to 2.17]
Statistical Analysis 3: Comparison: Tezepelumab vs Placebo; Influenza B Victoria Lineage Ratio of placebo over tezepelumab. Results based on ANCOVA model; Test type: Other; Geometric LS mean ratio = 1.23, 90% CI 2-sided [0.73 to 2.07]
Statistical Analysis 4: Comparison: Tezepelumab vs Placebo; Influenza B Yamagata Lineage Ratio of placebo over tezepelumab. Results based on ANCOVA model; Test type: Other; Geometeric LS mean ratio = 0.89, 90% CI 2-sided [0.54 to 1.48]

3. Primary Outcome: Post-vaccination Strain-specific Serum HAI Antibody Geometric Mean Titers (GMTs)
Description: as for outcome 1
Time Frame: Week 16
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Titer
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 33 | 33
Titer
  Influenza A H1N1 | 809.23 (0.921) [lower limit 0.921] | 596.76 (1.076) [lower limit 1.076]
  Influenza B Yamagata Lineage | 167.46 (0.925) [lower limit 0.925] | 161.56 (0.688) [lower limit 0.688]
  Influenza B Victoria Lineage | 194.68 (1.089) [lower limit 1.089] | 200.55 (0.948) [lower limit 0.948]
Statistical Analysis 1: Comparison: Tezepelumab vs Placebo; Influenza A H1N1 Ratio of placebo over tezepelumab. Results based on ANCOVA model; Test type: Other; Geometeric LS mean ratio = 0.74, 90% CI 2-sided [0.52 to 1.04]
Statistical Analysis 2: Comparison: Tezepelumab vs Placebo; Influenza B Yamagata Lineage Ratio of placebo over tezepelumab. Results based on ANCOVA model; Test type: Other; Geometeric LS mean ratio = 0.96, 90% CI 2-sided [0.72 to 1.29]
Statistical Analysis 3: Comparison: Tezepelumab vs Placebo; Influenza B Victoria Lineage Ratio of placebo over tezepelumab. Results based on ANCOVA model; Test type: Other; Geometric LS mean ratio = 1.03, 90% CI 2-sided [0.73 to 1.46]

4. Primary Outcome: Post-vaccination Strain-specific Serum MN Antibody GMTs
Description: as for outcome 2
Time Frame: Week 16
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Titer
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 33 | 33
Titer
  Influenza A H1N1 | 382.55 (1.469) [lower limit 1.469] | 303.63 (1.667) [lower limit 1.667]
  Influenza A H3N2 | 600.92 (2.154) [lower limit 2.154] | 457.33 (2.336) [lower limit 2.336]
  Influenza B Yamagata Lineage | 355.44 (1.076) [lower limit 1.076] | 366.81 (1.270) [lower limit 1.270]
  Influenza B Victoria Lineage | 125.67 (4.687) [lower limit 4.687] | 124.35 (3.515) [lower limit 3.515]
Statistical Analysis 1: Comparison: Tezepelumab vs Placebo; Influenza A H1N1 Ratio of placebo over tezepelumab. Results based on ANCOVA model; Test type: Other; Geometeric LS mean ratio = 0.79, 90% CI 2-sided [0.51 to 1.25]
Statistical Analysis 2: Comparison: Tezepelumab vs Placebo; Influenza A H3N2 Ratio of placebo over tezepelumab. Results based on ANCOVA model; Test type: Other; Geometeric LS mean ratio = 0.76, 90% CI 2-sided [0.42 to 1.28]
Statistical Analysis 3: Comparison: Tezepelumab vs Placebo; Influenza B Victoria Lineage Ratio of placebo over tezepelumab. Results based on ANCOVA model; Test type: Other; Geometric LS mean ratio = 0.99, 90% CI 2-sided [0.49 to 1.99]
Statistical Analysis 4: Comparison: Tezepelumab vs Placebo; Influenza B Yamagata Lineage Ratio of placebo over tezepelumab. Results based on ANCOVA model; Test type: Other; Geometeric LS mean ratio = 1.03, 90% CI 2-sided [0.70 to 1.52]

5. Primary Outcome: Percentage of Patients With Post-vaccination Strain-specific Antibody Response at Week 16 With Antibody Response Defined as a ≥ 4-fold Rise in HAI Antibody Titer
Description: as for outcome 1
Time Frame: Week 16
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 33 | 33
Percentage of participants
  Influenza A H1N1 | 78.8 (63.82) [63.82 to 89.60] | 51.5 (36.07) [36.07 to 66.74]
  Influenza B Yamagata Lineage | 15.2 (6.17) [6.17 to 29.25] | 15.2 (6.17) [6.17 to 29.25]
  Influenza B Victoria Lineage | 30.3 (17.46) [17.46 to 45.96] | 39.4 (25.11) [25.11 to 55.18]

6. Primary Outcome: Percentage of Patients With Post-vaccination Strain-specific Antibody Response at Week 16 With Antibody Response Defined as a ≥ 4-fold Rise in MN Antibody Titer
Description: Effect of tezepelumab on the humoral immune response following seasonal influenza virus vaccination in adolescent and young adult participants with moderate to severe asthma was assessed.
  Vaccine immunogenicity analysis set consisted of all randomised patients who received the influenza vaccine plus at least 1 dose of tezepelumab or placebo, had pre and post vaccination HAI or MN antibody measurements, had no influenza infection prior to Visit 7 (Week 16), and had no protocol deviation, judged to have the potential to interfere with the generation or interpretation of an antibody response.
Time Frame: Week 16
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 33 | 33
Percentage of participants
  Influenza A H1N1 | 81.8 (67.24) [67.24 to 91.77] | 75.8 (60.49) [60.49 to 87.32]
  Influenza A H3N2 | 60.6 (44.82) [44.82 to 74.89] | 51.5 (36.07) [36.07 to 66.74]
  Influenza B Yamagata Lineage | 51.5 (36.07) [36.07 to 66.74] | 36.4 (22.50) [22.50 to 52.16]
  Influenza B Victoria Lineage | 54.5 (38.94) [38.94 to 69.51] | 63.6 (47.84) [47.84 to 77.50]

7. Primary Outcome: Percentage of Patients With Post-vaccination Strain-specific HAI Antibody Titer ≥ 40
Description: as for outcome 1
Time Frame: Week 16
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 33 | 33
Percentage of participants
  Influenza A H1N1 | 100 (91.32) [91.32 to 100.00] | 100 (91.32) [91.32 to 100.00]
  Influenza B Yamagata Lineage | 97 (86.41) [86.41 to 99.84] | 100 (91.32) [91.32 to 100.00]
  Influenza B Victoria Lineage | 100 (91.32) [91.32 to 100.00] | 97.0 (86.41) [86.41 to 99.84]

8. Primary Outcome: Percentage of Patients With Post-vaccination Strain-specific MN Antibody Titer ≥ 40
Description: as for outcome 2
Time Frame: Week 16
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 33 | 33
Percentage of participants
  Influenza A H1N1 | 100 (91.32) [91.32 to 100.00] | 93.9 (82.13) [82.13 to 98.91]
  Influenza A H3N2 | 93.9 (82.13) [82.13 to 98.91] | 97 (86.41) [86.41 to 99.84]
  Influenza B Yamagata Lineage | 97 (86.41) [86.41 to 99.84] | 100 (91.32) [91.32 to 100.00]
  Influenza B Victoria Lineage | 78.8 (63.82) [63.82 to 89.60] | 81.8 (67.24) [67.24 to 91.77]

9. Secondary Outcome: Serum Tezepelumab Concentrations
Description: Tezepelumab serum concentrations were summarized using descriptive statistics at each visit.
Time Frame: Week 0, Week 12, Week 16 and Week 28
Population: Pharmacokinetic (PK) analysis set consisted of all patients who received tezepelumab and from whom PK blood samples were obtained and assumed not to be affected by factors such as protocol deviations.
  Here, Number of patients analyzed in each row reflects number of patients analyzed for that timepoint
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (μg/mL)
Arm/Group | Tezepelumab
Number analyzed (Participants) | 32
microgram/milliliter (μg/mL)
  Week 0 | NA (NA) — Not calculable as 31 of 32 participants had concentrations below lower limit of quantification (0.010 ug/ml). The remaining participant had serum concentration of 0.0235 ug/ml.
  Week 12: number analyzed (Participants) | 30
  Week 12 | 27.00 (0.5421)
  Week 16 | 20.76 (3.6969)
  Week 28: number analyzed (Participants) | 31
  Week 28 | 2.79 (1.0705)

10. Secondary Outcome: Immunogenicity
Description: Immunogenicity assessments were performed. ADA prevalence was defined as patients who are ADA positive at any time including baseline. Persistently positive was defined as having at least two post-baseline ADA positive measurements (with ≥16 weeks between first and last positive) or an ADA positive result at the last available post-baseline assessment. Transiently positive was defined as having at least one post-baseline ADA positive measurement and not fulfilling the conditions for persistently positive. Treatment boosted ADA was defined as baseline positive ADA titre that was boosted to a 4-fold or higher-level following treatment. Treatment emergent ADA (ADA incidence) was defined as the sum of treatment induced ADA and treatment boosted ADA.
Time Frame: From Baseline to Week 28
Population: Safety analysis set consisted of all patients who received at least 1 dose of study intervention.
Measure: Number; unit: Patients
Arm/Group | Tezepelumab | Placebo
Number analyzed (Participants) | 35 | 35
Patients
  ADA prevalence | 0 | 4
  Only baseline ADA positive | 0 | 0
  Both baseline and post-baseline ADA positive | 0 | 0
  Any baseline ADA positive | 0 | 0
  Any post-baseline ADA positive | 0 | 4
  Treatment-induced ADA positive | 0 | 4
  ADA persistently positive | 0 | 4
  ADA transiently positive | 0 | 0
  Treatment-boosted ADA positive | 0 | 0
  TE-ADA positive (ADA incidence) | 0 | 4

ADVERSE EVENTS:
Time Frame: From the date of the first dose of study drug, throughout the treatment period up to the follow-up period or end of the study visit (Week 28)
Arm/Group | Tezepelumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 1/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 1/35
Other Adverse Events (participants affected / at risk) | 14/35 | 15/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tezepelumab (N=35) | Placebo (N=35)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tezepelumab (N=35) | Placebo (N=35)
COVID-19 (Infections and infestations) | 8 (8) | 8 (8)
Acute sinusitis (Infections and infestations) | 3 (3) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains trade secrets and confidential commercial information, disclosure of which is prohibited without providing advance notice to AstraZeneca and opportunity to object.

DOCUMENTS (2):
  • Study Protocol (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/59/NCT05062759/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT05062759/SAP_001.pdf